CLINICAL TRIAL: NCT00992706
Title: Local Antiperspirant for Prevention of Palmar-Plantar Erythrodysesthesia (PPE) in Patients Treated With Pegylated Liposomal Doxorubicin: A Randomized, Multicenter, Double Blinded, Phase III Trial
Brief Title: F511 Cream in Preventing Palmar-Plantar Erythrodysesthesia in Patients Receiving Doxorubicin Hydrochloride Liposome for Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SAKK 92/08; SWS-SAKK-92/08; EU-20978; CDR0000652808
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer; Palmar-plantar Erythrodysesthesia
Keywords: palmar-plantar erythrodysesthesia; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hand-Foot Syndrome; Breast Neoplasms, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: antiperspirant cream F511 — Placebo and verum cream once daily, in the morning, during the first week of the first PLD treatment only, then once daily, three times per week (in the morning). Tube R for right hand and foot, tube L for left hand and foot.
Drug: pegylated liposomal doxorubicin hydrochloride — According to local practice. 1, 2 and 4 week schedules with at least 10mg/m2 per week are allowed.

SUMMARY:
RATIONALE: F511 cream may prevent or reduce palmar-plantar erythrodysesthesia in women receiving doxorubicin hydrochloride liposome for metastatic breast cancer.

PURPOSE: This randomized phase III trial is studying F511 cream to see how well it works compared with a placebo cream in preventing palmar-plantar erythrodysesthesia in patients receiving doxorubicin hydrochloride liposome for metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the effects of F511 cream on the occurrence of palmar-plantar erythrodysesthesia (PPE) in patients with metastatic breast cancer treated with pegylated liposomal doxorubicin hydrochloride.

OUTLINE: This is a multicenter study.

Patients receive pegylated liposomal doxorubicin hydrochloride according to local practice on 1, 2, or 4 weeks course schedules with at least 10 mg/m^2 per week allowed.

Patients apply F511 cream on one side, hand and foot and the corresponding placebo on the other side hand and foot once daily (the morning) during the first week of the first pegylated liposomal doxorubicin hydrochloride treatment only, then once daily, three times per week thereafter. Treatment continues throughout chemotherapy administration in the absence of palmar-plantar erythrodysesthesia (PPE) ≥ grade 2

After completion of study therapy, patients are followed for 30 days. Patients with PPE ≥ grade 2 are followed until the PPE resolves to ≤ grade 1.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic breast cancer

  * No cutaneous metastases on hands or feet
* Pegylated liposomal doxorubicin hydrochloride monotherapy is indicated according to the local investigator

  * Planned dose at least 10 mg/m^2 per week
* No sign of palmar-plantar erythrodysesthesia (PPE) at study entry

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Able to apply topical medication (cream) or provide for another person to apply cream
* Not pregnant or breastfeeding
* Fertile patients must use effective contraception during trial participation and for 1 month after completion
* Negative pregnancy test
* Compliant and geographically proximal in order to allow proper evaluation and follow-up
* No dermatologic conditions (e.g., psoriasis) that, in the opinion of the physician, may affect the hands or feet or may complicate evaluation during study treatment
* No known allergy or hypersensitivity to F511 cream

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 30 days since prior and no concurrent treatment with other experimental drugs or anticancer therapy
* More than 30 days since prior and no concurrent treatment on another clinical trial
* No concurrent local use of other ointments or creams for hands or feet other than Excipial Repair®

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Palmar-plantar erythrodysesthesia (PPE, hand-foot syndrome, HFS) grade ≥ 2 | Until PPE grade ≥2

SECONDARY OUTCOMES:
Patient-reported outcome | Until PPE grade ≥2
Adverse skin reaction to local therapy | Until PPE grade ≥2
Extent of symptom relief | Until PPE grade ≥2
Recurrence of PPE grade ≥ 2 | Until PPE grade ≥2

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ruhstaller, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (15):
- Switzerland (15):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Spitalzentrum Biel, Biel
  - Spital Buelach, Bülach
  - Kantonsspital Graubuenden, Chur
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Onkologie Schaffhausen, Schaffhausen
  - Institut Central des Hopitaux Valaisans, Sion
  - Kantonsspital Winterthur, Winterthur
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Templeton AJ, Ribi K, Surber C, Sun H, Hsu Schmitz SF, Beyeler M, Dietrich D, Borner M, Winkler A, Muller A, von Rohr L, Winterhalder RC, Rochlitz C, von Moos R, Zaman K, Thurlimann BJ, Ruhstaller T; Swiss Group for Clinical Cancer Research (SAKK) Coordinating Center. Prevention of palmar-plantar erythrodysesthesia with an antiperspirant in breast cancer patients treated with pegylated liposomal doxorubicin (SAKK 92/08). Breast. 2014 Jun;23(3):244-9. doi: 10.1016/j.breast.2014.02.005. Epub 2014 Mar 20. PMID 24656636